CLINICAL TRIAL: NCT06324565
Title: The Role of Preoperative D-dimer Levels in the Diagnosis of Adnexal Torsion in Children and Adolescents
Brief Title: Role of Preoperative D-dimer Levels in the Diagnosis of Adnexal Torsion
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 24/2021
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Adnexal Torsion
Keywords: D-dimer; Diagnosis; Adnexal torsion
MeSH Terms: conditions — Ovarian Torsion; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ovarian Torsion: All female patients under the age of 18 with suspicious signs and symptoms of ovarian torsion
  Interventions: Diagnostic Test: D-Dimer test

INTERVENTIONS:
Diagnostic Test: D-Dimer test — All patients in whom preoperative diagnostics have not been able to exclude a surgical pathology and who are candidates for diagnostic-therapeutic surgery will be referred for minimally invasive abdominal exploration in the real suspicion of ovarian torsion. During the pre-operative phase, blood exams will be performed including coagulation which will be integrated with the D-dimer values. In addition, as usual, the clinical examination of the patients will be performed integrated with the various diagnostic image tools generally used in this category of patients (abdomen ultrasound +/- magnetic resonance in urgency).

SUMMARY:
Adnexal torsion is the fifth most common gynecologic emergency. Thirty percent of all cases of adnexal torsion occur in females younger than 20 years. Approximately 5 of 100,000 females aged 1-20 years are affected, with girls older than 10 years at increased risk because of hormonal influences and gonadal growth that result in an increased frequency of physiologic and pathologic masses. The most common clinical symptom of torsion is sudden-onset abdominal pain that is intermittent, non-radiating, and associated with nausea and vomiting in 62% and 67% of cases respectively. Moreover, abdominal tenderness is a clinical sign which is reported in up to 88% of patients with adnexal torsion. None of the following tests are useful in the diagnosis of adnexal torsion: leukocytosis, pyuria, C-reactive protein, and erythrocyte sedimentation rate. Actually, transabdominal ultrasonography is the imaging modality of choice with a sensitivity of 92% and specificity of 96% in detecting adnexal torsion. A second-line imaging tool in the diagnosis of adnexal torsion is magnetic resonance, which may require a sedation in selected cases. Consequently, there are no clinical or imaging criteria sufficient to confirm the preoperative diagnosis of adnexal torsion to date. Therefore, patients with a clinical suspicion for adnexal torsion should undergo emergent diagnostic laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Age < 18 years
* presenting with lower quadrants abdominal pain
* Imaging suspicious for adnexal torsion

Exclusion Criteria:

* Female patients aged > 18 years
* Previous surgery for adnexal pathologies
* Clinical symptoms and imaging suggesting a different surgical pathology (i.e., appendicitis, gastroenteritis)

Max Age: 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Study Population: Girls younger than 18 years of age admitted to the Emergency Department for abdominal pain suspicious for adnexal torsion
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2024-12-13 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the D-Dimer | Through study completion, an average of 18 months
  Area under the Receiver Operating Characteristic (ROC) curve (AUC) will be assessed to evaluate the diagnostic accuracy of the D-Dimer

CONTACTS AND LOCATIONS:
Locations (9):
- Austria (2):
  - Medical University of Graz, Graz
  - Medical University of Vienna, Vienna
- Italy (5):
  - IRCCS Giannina Gaslini, Genova
  - Azienda Ospedale Università Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Presidio Ospedaliero Santa Chiara, Trento
  - Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste
- Serbia (2):
  - University of Belgrade, Belgrade
  - University of Novi Sad, Novi Sad